CLINICAL TRIAL: NCT06376708
Title: Comparison Between PEEK With Platelet-rich Fibrin and PEEK Alone in Maxillary Sinus Augmentation: Histomorphometric and Clinical Analysis: A Randomized Clinical Trial
Brief Title: Comparison Between PEEK With Platelet-rich Fibrin and PEEK Alone in Maxillary Sinus Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed gamal hammad, master holder, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-3-13
Record Dates: First submitted 2024-03-28; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-09

CONDITIONS: Maxillary Sinus
Keywords: maxillary sinus elevation and PEEK
MeSH Terms: interventions — polyetheretherketone

STUDY DESIGN:
Intervention Model Description: use of platelet rich fibrin after maxillary sinus elevation using PEEK
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEEK and PRF (Experimental): maxillary sinus elevation using PEEK and platelet rich fibrin
  Interventions: Other: platelet rich fibrin; Other: Polyether ether ketone
- PEEK alone (Active Comparator): maxillary sinus elevation using PEEK alone
  Interventions: Other: Polyether ether ketone

INTERVENTIONS:
Other: platelet rich fibrin — platelet rich fibrin
  Other Names: P.R.F
  Arms: PEEK and PRF
Other: Polyether ether ketone — Polyether ether ketone
  Other Names: PEEK

SUMMARY:
comparison between the resulted bone during maxillary sinus elevation by PEEK with and without platelet rich fibrin

DETAILED DESCRIPTION:
Histomorphometric and clinical analysis of the bone formed after 6 months after the maxillary sinus elevation using PEEK in the 2 groups : the study group (PEEK with platelet rich fibrin) and the control group (PEEK alone ) .

ELIGIBILITY:
Inclusion Criteria:

* • Posterior edentulous ridges with pneumatized maxillary sinus and remaining bone height less than 4 mm.

  * ASA physical status I and II.
  * Patients willing to be a part of the study and ready to give their consent in writing for the same.
  * Patient not complain from maxillary sinusitis
  * Patient with good oral hygiene.
  * Both males as well as females without any active periodontal disease.
  * The edentulous ridges are covered with optimal thickness of mucoperiosteum with no signs of inflammation, ulceration or scar tissue.
  * Remaining natural teeth have good periodontal tissue support and occlusion showed sufficient inter arch space for future prosthesis.

Exclusion Criteria:

* • General contraindications to implant surgery.

  * Untreated gingivitis, periodontitis.
  * Subjected to irradiation in the head and neck area less than 1 year before implantation.
  * Untreated periodontitis.
  * Pregnant or nursing.
  * Unable to open mouth sufficiently to accommodate the surgical tooling.
  * Patients participating in other studies, if the present protocol could not be properly followed.
  * Patient who could/would not participate in the follow-up period.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Bone quantity | 6 months postoperatively
  using of CBCT

SECONDARY OUTCOMES:
Bone quality | 6 months postoperatively
  Histomorphometic analysis (For Core biopsy)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No